CLINICAL TRIAL: NCT05007080
Title: A Randomized, Observer-blind, Phase 2 Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Different Dose Levels of Ad26.COV2.S Administered as a One- or Two-dose Regimen in Healthy Adolescents From 12 to 17 Years Inclusive
Brief Title: A Study to Evaluate Different Dose Levels of Ad26.COV2.S in Healthy Adolescents From 12 to 17 Years Inclusive
Acronym: HORIZON 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108966; 2020-005720-11 (EudraCT Number); VAC31518COV3006 (Other: Janssen Vaccines & Prevention B.V.)
Expanded Access: NCT04817657 (No longer available)
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Coronavirus Disease-2019 (COVID-19) Prevention
MeSH Terms: conditions — COVID-19 | interventions — Ad26COVS1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: Ad26.COV2.S Dose Level 1 (Lower Volume): 1-Dose Regimen (Experimental): Participants will receive 1-dose of Ad26.COV2.S at dose level 1 on Day 1 and placebo on Day 57. Participants will be unblinded to the primary vaccination regimen at 6 months after the first vaccination. Participants will receive booster vaccination at dose level 1 on Day 184.
  Interventions: Biological: Ad26.COV2.S
- Group 2: Ad26.COV2.S Dose Level 2: 1-Dose Regimen (Experimental): Participants will receive 1-dose of Ad26.COV2.S at dose level 2 on Day 1 and placebo on Day 57. Participants will be unblinded to the primary vaccination regimen at 6 months after the first vaccination. Participants will receive booster vaccination at dose level 1 on Day 184.
  Interventions: Biological: Ad26.COV2.S
- Group 3: Ad26.COV2.S Dose Level 3: 1-Dose Regimen (Experimental): Participants will receive 1-dose of Ad26.COV2.S at dose level 3 on Day 1 and placebo on Day 57. Participants will be unblinded to the primary vaccination regimen at 6 months after the first vaccination. Participants will receive booster vaccination at dose level 1 on Day 184.
  Interventions: Biological: Ad26.COV2.S
- Group 4: Ad26.COV2.S Dose Level 1: 2-Dose Regimen (Experimental): Participants will receive 2-dose of Ad26.COV2.S at dose level 1 on Day 1 and 57. Participants will be unblinded to the primary vaccination regimen at 6 months after the first vaccination.
  Interventions: Biological: Ad26.COV2.S
- Group 5: Ad26.COV2.S Dose Level 2: 2-Dose Regimen (Experimental): Participants will receive 2-doses of Ad26.COV2.S at dose level 2 on Day 1 and Day 57. Participants will be unblinded to the primary vaccination regimen at 6 months after the first vaccination.
  Interventions: Biological: Ad26.COV2.S
- Group 6: Ad26.COV2.S Dose Level 3: 2-Dose Regimen (Experimental): Participants will receive 2-doses of Ad26.COV2.S at dose level 3 on Day 1 and Day 57. Participants will be unblinded to the primary vaccination regimen at 6 months after the first vaccination.
  Interventions: Biological: Ad26.COV2.S

INTERVENTIONS:
Biological: Ad26.COV2.S — Ad26.COV2.S will be administered as intramuscular (IM) injection.
  Other Names: Ad26COVS1, VAC31518, JNJ-78436735

SUMMARY:
The primary purpose of this study is to assess the safety, reactogenicity, and humoral immune response of Ad26.COV2.S administered intramuscularly (IM) as a 1-dose schedule or as a 2-dose schedule (56-day interval) in adolescents.

DETAILED DESCRIPTION:
Available safety, immunogenicity and efficacy data from the Ad26.COV2.S vaccine development program supports initiating evaluation of Ad26.COV2.S in the pediatric population. Ad26.COV2.S will be evaluated in the pediatric population through a dose-confirmation approach. Ad26.COV2.S (also known as Ad26COVS1, VAC31518, JNJ-78436735) is a monovalent vaccine composed of a recombinant, replication-incompetent human adenovirus type 26 (Ad26) vector, constructed to encode the severe acute respiratory syndrome coronavirus(-2) (SARS-CoV-2) spike (S) protein, stabilized in its prefusion conformation. The study duration from screening until the last follow-up visit will be, excluding the 28-day screening phase, 8 months (Groups 4-6) to 12 months (Groups 1-3), consisting of 12-month study duration comprising a study period (6-months) including vaccination with a 1 active dose and a placebo vaccination (56-day interval), followed by a booster vaccination at 6 months and follow-up (safety and immunogenicity) until at least 6 months after booster vaccination (Groups 1-3) and 8 month study duration comprising 2 active doses (56-day interval) and follow-up (safety and immunogenicity) until at least 6 months after second vaccination (Groups 4-6). Assessments like immunogenicity (such as humoral and cellular immune responses), safety and reactogenicity (such as adverse events [AEs] monitoring) will be performed in this study. Other safety assessments include vital signs measurements (heart rate, supine systolic and diastolic blood pressure, respiratory rate, and body temperature) and physical examinations. The overall study duration from enrolment of the first participant until study completion is expected to be up to 1 year 11 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant's age is 12 to 17 years of age at the time of first vaccination
* Participant must be healthy, in the investigator's clinical judgement, as confirmed by medical history, physical examination, and vital signs performed at screening, and must not have comorbidities related to an increased risk of severe coronavirus disease-2019 (COVID-19)
* Participant agrees to not donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after receiving the last dose of study vaccine
* Participant and/or parent(s)/legal guardian(s) are available and willing to participate for the duration of the study visits and follow-up
* Each participant or participant's parent(s)/legal guardian(s) must have access to a consistent means of contact either by telephone contact or email/computer

Exclusion Criteria:

* Participant has a history of malignancy, bone marrow transplant, or solid organ transplant within 5 years before screening
* Participant has a known or suspected allergy, history of anaphylaxis, or other serious adverse reactions, related to vaccines or their excipients (including specifically the excipients of the study vaccine)
* Use of systemic corticosteroids at an immunosuppressive dose (treatment duration more than 14 days for one course or recurrent use) within 6 months before administration of study vaccine and during the study
* Participants with a history of illness or with an ongoing illness that, in the opinion of the investigator, may pose additional risk to the participant if he/she participates in the study
* Any serious, chronic, or progressive disease (example: diabetes, cardiac disease, hepatic disease, progressive neurological disease or seizure disorder; autoimmune disease, acquired immunodeficiency syndrome [AIDS] infection, blood dyscrasias, bleeding diathesis, signs of cardiac or renal failure, or severe malnutrition)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (18):
- Argentina (3):
  - CIPREC, Buenos Aires
  - Hospital de Ninos de Cordoba, Córdoba
  - Hospital del Niño Jesús, San Miguel de Tucumán
- Brazil (4):
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - CPQuali Pesquisa Clinica LTDA ME, São Paulo
- India (4):
  - Sri ramchandra Medical College & Research Institute, Chennai
  - JSS Hospital, Mysore
  - Supe Heart And Diabetes Hospital and Research Center, Nashik
  - BAPS Pramukhswami Hospital, Surat
- Mexico (2):
  - CAIMED Investigacion en salud S.A de C.V., Mexico City
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
- South Africa (5):
  - Ndlovu Elandsdoorn Site, Dennilton
  - Shandukani Research Centre, Johannesburg
  - Setshaba Research Centre, Soshanguve
  - Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital, Soweto
  - University of Witwatersrand - Helen Joseph Hospital - Themba Lethu Hiv Research Centre, Westdene Johannesburg Gauteng

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Tica J, Rezelj VV, Baron B, van Paassen V, Zaidman J, Fairlie L, Scheper G, Le Gars M, Struyf F, Douoguih M, Ruiz-Guinazu J; COV3006 study group; COV3006 Study Group Collaborators. Safety and immunogenicity of Ad26.COV2.S in adolescents: Phase 2 randomized clinical trial. Hum Vaccin Immunother. 2025 Dec;21(1):2450120. doi: 10.1080/21645515.2025.2450120. Epub 2025 Jan 27. PMID 39868766

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 304 randomized participants, 3 participants were randomized to an arm that was closed prior to vaccination due to ethical reasons. One participant was excluded from the analysis due to lack of a valid informed consent form and is not presented in the below table.
Groups:
- Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo: Participants received a single dose of Ad26.COV.S 2.5*10^10 virus particle (vp) as intramuscular (IM) injection on Day 1 and placebo matching to Ad26.COV.S 2.5*10^10 vp as IM injection on Day 57. Participants were unblinded to the primary vaccination regimen at 6 months after the first vaccination. Participants received booster vaccination with Ad26.COV.S 2.5*10^10 vp on Day 184.
- Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo: Participants received a single dose of Ad26.COV2.S 1.25*10^10 vp as IM injection on Day 1 and placebo matching to Ad26.COV2.S 1.25*10^10 vp as IM injectionon Day 57. Participants were unblinded to the primary vaccination regimen at 6 months after the first vaccination. Participants received booster vaccination with Ad26.COV.S 2.5*10^10 vp on Day 184.
- Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo: Participants received a single dose of Ad26.COV2.S 0.625*10^10 vp as IM injection on Day 1 and placebo matching to Ad26.COV2.S 0.625*10^10 vp as IM injection Day 57. Participants were unblinded to the primary vaccination regimen at 6 months after the first vaccination. Participants received booster vaccination with Ad26.COV.S 2.5*10^10 vp on Day 184.
- Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp: Participants received a single dose of Ad26.COV2.S 2.5*10^10 vp as IM injection on Day 1 and Day 57. Participants were unblinded to the primary vaccination regimen at 6 months after the first vaccination.
- Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp: Participants received a single dose of Ad26.COV2.S 1.25*10^10 vp as IM injection on Day 1 and Day 57. Participants were unblinded to the primary vaccination regimen at 6 months after the first vaccination
- Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp: Participants received a single dose of Ad26.COV2.S 0.625*10^10 vp as IM injection on Day 1 and Day 57. Participants were unblinded to the primary vaccination regimen at 6 months after the first vaccination.
Period: Overall Study
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Started | 51 | 50 | 51 | 49 | 49 | 50
Vaccinated | 51 | 50 | 51 | 49 | 49 | 49
Completed | 49 | 46 | 50 | 45 | 47 | 45
Not Completed | 2 | 4 | 1 | 4 | 2 | 5
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 1 | 1
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 2 | 1 | 1
Not completed — Other | 1 | 0 | 1 | 1 | 0 | 2
Not completed — Randomized not vaccinated | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants with at least one vaccine administration documented.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp | Total
Number analyzed (Participants) | 51 | 50 | 51 | 49 | 49 | 49 | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.87) | 14 (1.82) | 14.3 (1.76) | 14.4 (1.75) | 14.2 (1.8) | 14.1 (1.84) | 14.2 (1.80)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adolescents (12-17 years) | 51 | 50 | 51 | 49 | 49 | 49 | 299
  Adults (18-64 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  From 65 to 84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 21 | 20 | 21 | 20 | 126
  Male | 29 | 28 | 30 | 29 | 28 | 29 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 19 | 24 | 17 | 16 | 26 | 124
  Not Hispanic or Latino | 29 | 30 | 27 | 32 | 31 | 23 | 172
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 1 | 0 | 2 | 2 | 12
  Asian | 17 | 19 | 17 | 22 | 19 | 14 | 108
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 17 | 13 | 16 | 12 | 14 | 16 | 88
  White | 13 | 13 | 14 | 12 | 13 | 17 | 82
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 3 | 2 | 1 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Groups 1, 2, 3, 4, 5 and 6: Number of Participants With Solicited Local Adverse Events (AEs) at 7 Days Post-dose 1
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited AEs were used to assess the reactogenicity of the study vaccine and were pre-defined as local (at the injection site) AEs for which participants were specifically asked and which were noted by participants in their reactogenicity diary for 7 days post each vaccination. Solicited local AEs are: injection site pain/tenderness, erythema, swelling at the vaccination site.
Time Frame: 7 days post-dose 1 on Day 1 (Day 8)
Population: Safety analyses set included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo: Participants received a single dose of Ad26.COV.S 2.5*10^10 vp as IM injection on Day 1 and placebo matching to Ad26.COV.S 2.5*10^10 vp as IM injection on Day 57. Participants were unblinded to the primary vaccination regimen at 6 months after the first vaccination. Participants received booster vaccination with Ad26.COV.S 2.5*10^10 vp on Day 184.
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 51 | 50 | 51 | 49 | 49 | 49
Participants | 13 | 16 | 17 | 11 | 12 | 15

2. Primary Outcome: Groups 1, 2, 3, 4, 5 and 6: Number of Participants With Solicited Local Adverse Events (AEs) at 7 Days Post-dose 2
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited AEs were used to assess the reactogenicity of the study vaccine and were pre-defined as local (at the injection site) AEs for which participants were specifically asked and which were noted by participants in their reactogenicity diary for 7 days post each vaccination. Solicited local AEs were: injection site pain/tenderness, erythema, swelling at the vaccination site.
Time Frame: 7 days post-dose 2 on Day 57 (Day 64)
Population: Safety analyses set included all participants with at least one vaccine administration documented. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp: Participants received single doses of Ad26.COV2.S 2.5*10^10 vp as IM injection on Day 1 and Day 57. Participants were unblinded to the primary vaccination regimen at 6 months after the first vaccination.
- Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp: Participants received single doses of Ad26.COV2.S 1.25*10^10 vp as IM injection on Day 1 and Day 57. Participants were unblinded to the primary vaccination regimen at 6 months after the first vaccination
- Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp: Participants received single doses of Ad26.COV2.S 0.625*10^10 vp as IM injection on Day 1 and Day 57. Participants were unblinded to the primary vaccination regimen at 6 months after the first vaccination.
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 51 | 50 | 50 | 47 | 49 | 48
Participants | 8 | 10 | 3 | 16 | 9 | 10

3. Primary Outcome: Groups 1, 2, 3, 4, 5 and 6: Number of Participants With Solicited Systemic AEs at 7 Days Post-dose 1
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited AEs were used to assess the reactogenicity of the study vaccine and were predefined as systemic AES for which participants were specifically asked and which were noted by participants in their reactogenicity diary for 7 days post each vaccination. Participants were instructed on how to note signs and symptoms in the diary on a daily basis for 7 days post-vaccination (day of vaccination and the subsequent 7 days) for the following solicited systemic AEs: fatigue, headache, nausea, myalgia and pyrexia.
Time Frame: 7 days post-dose 1 on Day 1 (Day 8)
Population: Safety analyses set included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 51 | 50 | 51 | 49 | 49 | 49
Participants | 20 | 13 | 18 | 14 | 16 | 16

4. Primary Outcome: Groups 1, 2, 3, 4, 5 and 6: Number of Participants With Solicited Systemic AEs at 7 Days Post-dose 2
Description: as for outcome 3
Time Frame: 7 days post-dose 2 on Day 57 (Day 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 51 | 50 | 50 | 47 | 49 | 48
Participants | 11 | 10 | 4 | 14 | 10 | 11

5. Primary Outcome: Groups 1, 2, 3, 4, 5 and 6: Number of Participants With Unsolicited AEs at 28 Days Post-dose 1
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited AEs that started within 7 days after vaccination but were ongoing after this 7-day window after each vaccination are also considered unsolicited AEs. Unsolicited AEs were defined as AEs for which the participants were not specifically questioned in the participant's reactogenicity diary.
Time Frame: 28 days post-dose 1 on Day 1 (Day 29)
Population: Safety analyses set included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 51 | 50 | 51 | 49 | 49 | 49
Participants | 9 | 9 | 5 | 3 | 8 | 10

6. Primary Outcome: Groups 1, 2, 3, 4, 5 and 6: Number of Participants With Unsolicited AEs at 28 Days Post-dose 2
Description: Description:
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited AEs that started within 7 days after vaccination but were ongoing after this 7-day window after each vaccination are also considered unsolicited AEs. Unsolicited AEs were defined as AEs for which the participants were not specifically questioned in the participant's reactogenicity diary.
Time Frame: 28 days post-dose 2 on Day 57 (Day 85)
Population: Safety analyses set included all participants with at least one vaccine administration documented. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure and "n" (number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 51 | 50 | 50 | 47 | 49 | 48
Participants | 7 | 7 | 8 | 7 | 7 | 9

7. Primary Outcome: Groups 1, 2, 3, 4, and 5: Number of Participants With Medically-attended Adverse Events (MAAEs) 6 Months Post-Dose 1
Description: MAAEs were defined as AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Routine study visits were not be considered medically-attended visits. New onset of chronic diseases were collected as part of the MAAEs.
Time Frame: From the first vaccination (Day 1) until 6 months post-dose 1 on Day 1 (Up to Day 184)
Population: Safety analyses set included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 51 | 50 | 51 | 49 | 49 | 49
Participants | 2 | 0 | 0 | 1 | 0 | 5

8. Primary Outcome: Groups 1, 2, 3, 4, 5 and 6: Number of Participants With MAAEs 6 Months Post-Dose 2
Description: as for outcome 7
Time Frame: From the first vaccination (Day 1) until 6 months post-dose 2 on Day 57 (Up to Day 240)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 51 | 50 | 50 | 47 | 49 | 48
Participants | 4 | 6 | 2 | 2 | 4 | 5

9. Primary Outcome: Groups 1, 2, and 3: Number of Participants With MAAEs Leading to Discontinuation
Description: Number of participants with MAAEs leading to discontinuation were reported. MAAEs were defined as AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Routine study visits were not be considered medically-attended visits. New onset of chronic diseases were collected as part of the MAAEs.
Time Frame: From first vaccination on Day 1 up to Day 366 (6 months after booster vaccination on Day 184)
Population: Safety analyses set included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo
Number analyzed (Participants) | 51 | 50 | 51
Participants | 0 | 0 | 0

10. Primary Outcome: Groups 4, 5 and 6: Number of Participants With MAAEs Leading to Discontinuation
Description: as for outcome 9
Time Frame: From first vaccination on Day 1 up to Day 240 (6 months after second vaccination on Day 57)
Population: Safety analyses set included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 49 | 49 | 49
Participants | 0 | 0 | 0

11. Primary Outcome: Groups 1, 2, and 3: Number of Participants With Serious Adverse Events (SAEs)
Description: SAE were defined as any untoward medical occurrence that at any dose results in any of the following outcomes: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Time Frame: From first vaccination on Day 1 up to Day 366 (6 months after booster vaccination on Day 184)
Population: Safety analyses set included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo
Number analyzed (Participants) | 51 | 50 | 51
Participants | 1 | 1 | 0

12. Primary Outcome: Groups 4, 5 and 6: Number of Participants With Serious Adverse Events (SAEs)
Description: as for outcome 11
Time Frame: From first vaccination on Day 1 up to Day 240 (6 months after second vaccination on Day 57)
Population: Safety analyses set included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 49 | 49 | 49
Participants | 0 | 1 | 0

13. Primary Outcome: Groups 1, 2, and 3: Number of Participants With Adverse Events of Special Interest (AESI) (Including Multisystem Inflammatory Syndrome in Children [MIS-C])
Description: Number of participants with AESI (including MIS-C) were reported. Thrombotic events (suspected deep vessel venous or arterial thrombotic events); Thrombocytopenia (platelet count below 150,000/μL) and MIS-C (a subject <21 years with fever, evidence of inflammation, and evidence of clinically severe illness requiring hospitalization, with multisystem (≥2) organ involvement [cardiac, renal, respiratory, hematologic, gastrointestinal, dermatologic or neurological]; & No alternative diagnoses; & Positive for ositive for current or recent (SARS-CoV-2) coronavirus disease 2019 [COVID-19] infection by Real-time reverse transcriptase-polymerase chain reaction [RT-PCR], serology, or antigen test; Or COVID-19 exposure within the 4 weeks prior to the onset of symptoms) were considered AESIs in this study.
Time Frame: From first vaccination on Day 1 up to Day 366 (6 months after booster vaccination on Day 184)
Population: Safety analyses set included all participants with at least one vaccine administration documented. 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo
Number analyzed (Participants) | 13 | 18 | 15
Participants | 0 | 0 | 0

14. Primary Outcome: Groups 4, 5 and 6: Number of Participants With AESI (Including MIS-C)
Description: Number of participants with AESI (including MIS-C) were reported. Thrombotic events: suspected deep vessel venous or arterial thrombotic events and Thrombocytopenia, defined as platelet count below 150,000/μL and MIS-C were considered as AESIs in this study. MIS-C, defined as: An individual aged <21 years presenting with fever, laboratory evidence of inflammation, and evidence of clinically severe illness requiring hospitalization, with multisystem (≥2) organ involvement (cardiac, renal, respiratory, hematologic, gastrointestinal, dermatologic,or neurological); AND No alternative plausible diagnoses; AND Positive for current or recent SARS-CoV-2 (COVID-19) infection by RT-PCR, serology, or antigen test; or COVID-19 exposure within the 4 weeks prior to the onset of symptoms.
Time Frame: From first vaccination on Day 1 up to Day 240 (6 months after second vaccination on Day 57)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 46 | 47 | 47
Participants | 0 | 0 | 0

15. Primary Outcome: Groups 1, 2, 3, 4, 5 and 6: Serological Response to Vaccination Measured by Spike-enzyme-linked Immunosorbent Assay (S-ELISA) at 28 Days Post-dose 1
Description: Serological response to vaccination measured by S-ELISA (ELISA Unit/milliliter (EU/mL)) at 28 days post-dose 1 were reported. For Vaccine-specific responses, a participant was defined as a responder if: 1. a baseline sample value of less than or equal to the lower limit of quantification (<=LLOQ) and a postbaseline sample strictly greater than the LLOQ; or 2. a baseline sample value strictly >LLOQ and a postbaseline sample value representing an at least 4-fold increase from the baseline sample value, was reported.
Time Frame: 28 days post-dose 1 on Day 1 (Day 29)
Population: The Per Protocol Immunogenicity (PPI) set included all randomized and vaccinated participants for whom immunogenicity data were available excluding data from participants with major protocol deviations expected to impact the immunogenicity outcomes. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Unit/milliliter (EU/mL)
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 44 | 42 | 43 | 35 | 39 | 41
ELISA Unit/milliliter (EU/mL) | 6533 (4341) [4341 to 9831] | 7812 (5120) [5120 to 11920] | 5881 (3719) [3719 to 9302] | 9273 (5596) [5596 to 15366] | 6758 (4344) [4344 to 10513] | 6069 (3780) [3780 to 9745]

16. Primary Outcome: Groups 1, 2, 3, 4, 5 and 6: Serological Response to Vaccination Measured by S-ELISA at 14 Days Post-dose 2
Description: Serological response to vaccination measured by S-ELISA (EU/mL) at 14 days post-dose 2 were reported. For Vaccine-specific responses, a participant was defined as a responder if: 1. a baseline sample value of <=LLOQ and a postbaseline sample strictly greater than the LLOQ; or 2. a baseline sample value strictly >LLOQ and a postbaseline sample value representing an at least 4-fold increase from the baseline sample value, was reported.
Time Frame: 14 days post-dose 2 on Day 57 (Day 71)
Population: The PPI set included all randomized and vaccinated participants for whom immunogenicity data were available excluding data from participants with major protocol deviations expected to impact the immunogenicity outcomes. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 38 | 31 | 38 | 30 | 32 | 37
EU/mL | 4923 (3329) [3329 to 7282] | 4679 (2748) [2748 to 7967] | 4043 (2480) [2480 to 6590] | 8958 (6333) [6333 to 12671] | 8716 (6577) [6577 to 11550] | 6522 (4461) [4461 to 9533]

17. Primary Outcome: Groups 1, 2, 3, 4, 5 and 6: Serological Response to Vaccination Measured by Virus Neutralization Assay (VNA) Titers 28 Days Post-dose 1
Description: Serological response to vaccination measured by VNA titers at 28 days post-dose 1 were reported. For Vaccine-specific responses, a participant was defined as a responder if: 1. a baseline sample value of <=LLOQ and a postbaseline sample strictly greater than the LLOQ; or 2. a baseline sample value strictly >LLOQ and a postbaseline sample value representing an at least 4-fold increase from the baseline sample value, was reported. Data were expressed as 50 percent (%) inhibitory concentration (IC50) units.
Time Frame: 28 days post-dose 1 on Day 1 (Day 29)
Population: The PPI set included all randomized and vaccinated participants for whom immunogenicity data were available excluding data from participants with major protocol deviations expected to impact the immunogenicity outcomes. Here "N" number of participants analyzed signifies the number of participants that were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 43 | 42 | 42 | 35 | 39 | 41
Titers | 1325 [792 to 2216] | 1754 [988 to 3113] | 1392 [806 to 2403] | 2038 [1065 to 3897] | 1878 [1089 to 3240] | 1455 [864 to 2449]

18. Primary Outcome: Serological Response to Vaccination Measured by VNA Titers 14 Days Post-dose 2
Description: Serological response to vaccination measured by VNA titers 14 days post-dose 2 were reported. For Vaccine-specific responses, a participant was defined as a responder if: 1. a baseline sample value of <=LLOQ and a postbaseline sample strictly greater than the LLOQ; or 2. a baseline sample value strictly >LLOQ and a postbaseline sample value representing an at least 4-fold increase from the baseline sample value, was reported. Data were expressed as IC50 units.
Time Frame: 14 days post-dose 2 on Day 57 (Day 71)
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 38 | 31 | 38 | 30 | 32 | 37
Titers | 1187 [698 to 2018] | 1094 [517 to 2315] | 864 [471 to 1583] | 2386 [1453 to 3917] | 2670 [1816 to 3925] | 1742 [1064 to 2852]

19. Secondary Outcome: Groups 1, 2, 3, 4, 5 and 6: Serological Response to Vaccination Measured by Binding Antibody Titers to Severe Acute Respiratory Syndrome Coronavirus(-2) (SARS-CoV-2) or Individual SARS-CoV-2 S Proteins as Assessed by ELISA
Description: Serological response to vaccination measured by binding antibody titers to SARS-CoV-2 or individual SARS-CoV-2 S proteins as assessed by ELISA were reported. For Vaccine-specific responses, a participant was defined as a responder if: 1. a baseline sample value of <=LLOQ and a postbaseline sample strictly greater than the LLOQ; or 2. a baseline sample value strictly >LLOQ and a postbaseline sample value representing an at least 4-fold increase from the baseline sample value, was reported.
Time Frame: Groups 1-3: Days 1, 29, 57, 71, 184, 198, and 366; Groups 4-6: Days 1, 29, 57, 71 and 240
Population: PPI set: all randomized and vaccinated participants with available immunogenicity data excluding data from participants with major protocol deviations expected to impact immunogenicity outcomes. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure, and "n"(number analyzed) signifies participants analyzed at specified timepoints (where "n=0", data were not planned to be analyzed at specified timepoint for specific arm).
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 51 | 50 | 51 | 49 | 49 | 49
EU/mL
  Day 1: number analyzed (Participants) | 51 | 50 | 51 | 49 | 48 | 49
  Day 1 | 255 [148 to 438] | 297 [156 to 563] | 338 [189 to 605] | 256 [144 to 455] | 200 [117 to 341] | 282 [151 to 528]
  Day 29: number analyzed (Participants) | 44 | 42 | 43 | 35 | 39 | 41
  Day 29 | 6533 [4341 to 9831] | 7812 [5120 to 11920] | 5881 [3719 to 9302] | 9273 [5596 to 15366] | 6758 [4344 to 10513] | 6069 [3780 to 9745]
  Day 57: number analyzed (Participants) | 41 | 40 | 41 | 33 | 38 | 38
  Day 57 | 5629 [3896 to 8133] | 7450 [4934 to 11249] | 4554 [2922 to 7099] | 7034 [4542 to 10891] | 5650 [3798 to 8405] | 4817 [3009 to 7710]
  Day 71: number analyzed (Participants) | 38 | 31 | 38 | 30 | 32 | 37
  Day 71 | 4923 [3329 to 7282] | 4679 [2748 to 7967] | 4043 [2480 to 6590] | 8958 [6333 to 12671] | 8716 [6577 to 11550] | 6522 [4461 to 9533]
  Day 184: number analyzed (Participants) | 19 | 11 | 19 | 0 | 0 | 0
  Day 184 | 4131 [2431 to 7021] | 4765 [2048 to 11087] | 3861 [1826 to 8165] |  |  |
  Day 198: number analyzed (Participants) | 27 | 21 | 31 | 0 | 0 | 0
  Day 198 | 6782 [5230 to 8795] | 7656 [5317 to 11026] | 10506 [8227 to 13417] |  |  |
  Day 240: number analyzed (Participants) | 0 | 0 | 0 | 14 | 16 | 22
  Day 240 |  |  |  | 4994 [3144 to 7932] | 5338 [3039 to 9377] | 3877 [2390 to 6289]
  Day 366: number analyzed (Participants) | 25 | 18 | 31 | 0 | 0 | 0
  Day 366 | 5087 [3809 to 6793] | 4934 [2856 to 8526] | 6585 [4907 to 8838] |  |  |

20. Secondary Outcome: Groups 1, 2, 3, 4, 5 and 6: Serological Response to Vaccination Measured by Neutralizing Antibody Titers to SARS-CoV-2
Description: Serological response to vaccination measured by neutralizing antibody titers to SARS-CoV-2 (VNA) were reported. For Vaccine-specific responses, a participant was defined as a responder if: 1. a baseline sample value of <=LLOQ and a postbaseline sample strictly greater than the LLOQ; or 2. a baseline sample value strictly >LLOQ and a postbaseline sample value representing an at least 4-fold increase from the baseline sample value, was reported. Data were expressed as IC50 units.
Time Frame: Groups 1-3: Days 1, 29, 57, 71, 184, 198 and 366; Groups 4-6: Days 1, 29, 57, 71 and 240
Population: PPI set: all randomized and vaccinated participants with available immunogenicity data excluding data from participants with major protocol deviations expected to impact immunogenicity outcomes. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure, and "n"(number analyzed) signifies participants analyzed at specified timepoints (where "n=0", data were not planned to be analyzed at specified timepoint for specific arm). "NA"=<LLOQ.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
Number analyzed (Participants) | 51 | 50 | 50 | 48 | 48 | 49
Titers
  Day 1 | 105 [NA to 163] — "NA" signifies that the value is <LLOQ. | 149 [88 to 250] | 114 [NA to 186] — "NA" signifies that the value is <LLOQ. | 112 [NA to 184] — "NA" signifies that the value is <LLOQ. | 83 [NA to 121] — "NA" signifies that the value is <LLOQ. | 127 [77 to 210]
  Day 29: number analyzed (Participants) | 43 | 42 | 42 | 35 | 39 | 41
  Day 29 | 1325 [792 to 2216] | 1754 [988 to 3113] | 1392 [806 to 2403] | 2038 [1065 to 3897] | 1878 [1089 to 3240] | 1455 [864 to 2449]
  Day 57: number analyzed (Participants) | 41 | 40 | 41 | 33 | 38 | 38
  Day 57 | 1197 [710 to 2020] | 1743 [992 to 3065] | 993 [570 to 1730] | 1662 [923 to 2992] | 1434 [847 to 2427] | 1188 [649 to 2173]
  Day 71: number analyzed (Participants) | 38 | 31 | 38 | 30 | 32 | 37
  Day 71 | 1187 [698 to 2018] | 1094 [517 to 2315] | 864 [471 to 1583] | 2386 [1453 to 3917] | 2670 [1816 to 3925] | 1742 [1064 to 2852]
  Day 184: number analyzed (Participants) | 19 | 11 | 19 | 0 | 0 | 0
  Day 184 | 1358 [773 to 2386] | 1702 [462 to 6273] | 860 [326 to 2267] |  |  |
  Day 198: number analyzed (Participants) | 27 | 21 | 31 | 0 | 0 | 0
  Day 198 | 2496 [1760 to 3539] | 2547 [1223 to 5303] | 4083 [3006 to 5547] |  |  |
  Day 240: number analyzed (Participants) | 0 | 0 | 0 | 14 | 16 | 22
  Day 240 |  |  |  | 1867 [944 to 3692] | 1900 [1035 to 3489] | 1134 [548 to 2347]
  Day 366: number analyzed (Participants) | 25 | 18 | 31 | 0 | 0 | 0
  Day 366 | 1809 [1231 to 2656] | 1783 [691 to 4599] | 2274 [1521 to 3401] |  |  |

21. Secondary Outcome: Groups 1, 2 and 3: Number of Participants With Solicited Local AEs for 7 Days Post-booster Vaccination
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited AEs were used to assess the reactogenicity of the study vaccine and were pre-defined as local (at the injection site) AEs for which participants were specifically asked and which were noted by participants in their reactogenicity diary for 7 days post each vaccination. Solicited local AEs are: injection site pain/tenderness, erythema, swelling at the vaccination site. Data for this outcome measure was not planned to be collected and analyzed for groups 4, 5 and 6 as pre-specified in the study protocol.
Time Frame: From first vaccination on Day 1 up to Day 191 (7 days after booster vaccination on Day 184)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo
Number analyzed (Participants) | 51 | 48 | 49
Participants | 19 | 16 | 17

22. Secondary Outcome: Groups 1, 2 and 3: Number of Participants With Solicited Systemic AEs for 7 Days Post-booster Vaccination
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited AEs were used to assess the reactogenicity of the study vaccine and were predefined as systemic AES for which participants were specifically asked and which were noted by participants in their reactogenicity diary for 7 days post each vaccination. Participants were instructed on how to note signs and symptoms in the diary on a daily basis for 7 days post-vaccination (day of vaccination and the subsequent 7 days) for the following solicited systemic AEs: fatigue, headache, nausea, myalgia and pyrexia. Data for this outcome measure was not planned to be collected and analyzed for groups 4, 5 and 6 as pre-specified in the study protocol.
Time Frame: From first vaccination on Day 1 up to Day 191 (7 days after booster vaccination on Day 184)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo
Number analyzed (Participants) | 51 | 48 | 49
Participants | 16 | 14 | 15

23. Secondary Outcome: Groups 1, 2 and 3: Number of Participants With Unsolicited AEs for 28 Days Post-booster Vaccination
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited AEs that started within 7 days after vaccination but were ongoing after this 7-day window after each vaccination are also considered unsolicited AEs. Unsolicited AEs were defined as AEs for which the participants were not specifically questioned in the participant's reactogenicity diary. Data for this outcome measure was not planned to be collected and analyzed for groups 4, 5 and 6 as pre-specified in the study protocol.
Time Frame: From first vaccination on Day 1 up to Day 212 (28 days after booster Vaccination on Day 184)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo
Number analyzed (Participants) | 51 | 48 | 49
Participants | 6 | 8 | 10

24. Secondary Outcome: Groups 1, 2 and 3: Number of Participants With MAAEs Until 6 Months Post-booster Vaccination
Description: MAAEs were defined as AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Routine study visits were not be considered medically-attended visits. New onset of chronic diseases were collected as part of the MAAEs. Data for this outcome measure was not planned to be collected and analyzed for groups 4, 5 and 6 as pre-specified in the study protocol.
Time Frame: From first vaccination on Day 1 up to Day 366 (6 months after booster vaccination on Day 184)
Population: Safety analyses set included all participants with at least one vaccine administration documented. Here, 'N' (number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo
Number analyzed (Participants) | 51 | 48 | 49
Participants | 1 | 2 | 2

25. Secondary Outcome: Groups 1, 2 and 3: Serological Response to Post-booster Vaccination Measured by Binding (S-ELISA) Antibody Titers
Description: Serological response to post-booster vaccination measured by binding (S-ELISA) antibody titers were reported. For Vaccine-specific responses, a participant was defined as a responder if: 1. a baseline sample value of <=LLOQ and a postbaseline sample strictly greater than the LLOQ; or 2. a baseline sample value strictly >LLOQ and a postbaseline sample value representing an at least 4-fold increase from the baseline sample value, was reported. Data for this outcome measure was not planned to be collected and analyzed for groups 4, 5 and 6 as pre-specified in protocol.
Time Frame: Days 184, 198 and 366
Population: PPI set: All randomized and vaccinated participants with available immunogenicity data excluding data from participants with major protocol deviations expected to impact the immunogenicity outcomes. Here, 'N' (number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure and "n" (number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo
Number analyzed (Participants) | 27 | 21 | 31
EU/mL
  Day 184: number analyzed (Participants) | 19 | 11 | 19
  Day 184 | 4131 [2431 to 7021] | 4765 [2048 to 11087] | 3861 [1826 to 8165]
  Day 198 | 6782 [5230 to 8795] | 7656 [5317 to 11026] | 10506 [8227 to 13417]
  Day 366: number analyzed (Participants) | 25 | 18 | 31
  Day 366 | 5087 [3809 to 6793] | 4934 [2856 to 8526] | 6585 [4907 to 8838]

26. Secondary Outcome: Groups 1, 2 and 3: Serological Response to Post-booster Vaccination Measured by Neutralizing (VNA) Antibody Titers
Description: Serological response to post-booster vaccination measured by neutralizing (VNA) antibody titers were reported. For Vaccine-specific responses, a participant was defined as a responder if: 1. a baseline sample value of <=LLOQ and a postbaseline sample strictly greater than the LLOQ; or 2. a baseline sample value strictly >LLOQ and a postbaseline sample value representing an at least 4-fold increase from the baseline sample value, was reported. Data were expressed as IC50 units. Data for this outcome measure was not planned to be collected and analyzed for groups 4, 5 and 6 as pre-specified in protocol.
Time Frame: Days 184, 198 and 366
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo
Number analyzed (Participants) | 27 | 21 | 31
Titers
  Day 184: number analyzed (Participants) | 19 | 11 | 19
  Day 184 | 1358 [773 to 2386] | 1702 [462 to 6273] | 860 [326 to 2267]
  Day 198 | 2496 [1760 to 3539] | 2547 [1223 to 5303] | 4083 [3006 to 5547]
  Day 366: number analyzed (Participants) | 25 | 18 | 31
  Day 366 | 1809 [1231 to 2656] | 1783 [691 to 4599] | 2274 [1521 to 3401]

ADVERSE EVENTS:
Time Frame: Groups 1, 2, 3: From first vaccination on Day 1 untill 6 months after booster vaccination on Day 184 (end of study) (up to Day 366) Groups 4, 5, 6: From first vaccination on Day 1 until 6 months after second vaccination on Day 57 (end of study) (up to Day 240)
Description: Safety analyses included all subjects with at least one vaccine administration documented.
Arm/Group | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/50 | 0/51 | 0/49 | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/51 | 1/50 | 0/51 | 0/49 | 1/49 | 0/49
Other Adverse Events (participants affected / at risk) | 35/51 | 32/50 | 34/51 | 26/49 | 29/49 | 35/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo (N=51) | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo (N=50) | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo (N=51) | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp (N=49) | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp (N=49) | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp (N=49)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal Cyst Excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ad26.COV2.S 2.5*10^10 vp + Placebo (N=51) | Group 2: Ad26.COV2.S 1.25*10^10 vp + Placebo (N=50) | Group 3: Ad26.COV2.S 0.625*10^10 vp + Placebo (N=51) | Group 4: Ad26.COV2.S 2.5*10^10 vp + Ad26.COV2.S 2.5*10^10 vp (N=49) | Group 5: Ad26.COV2.S 1.25*10^10 vp + Ad26.COV2.S 1.25*10^10 vp (N=49) | Group 6: Ad26.COV2.S 0.625*10^10 vp + Ad26.COV2.S 0.625*10^10 vp (N=49)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nausea(Solicited) (Gastrointestinal disorders) | 8 (8) | 5 (6) | 11 (13) | 6 (7) | 7 (8) | 2 (3)
Fatigue(Solicited) (General disorders) | 20 (26) | 11 (17) | 12 (14) | 16 (21) | 10 (11) | 14 (16)
Pyrexia(Solicited) (General disorders) | 10 (12) | 2 (4) | 7 (7) | 7 (7) | 2 (2) | 5 (5)
Vaccination Site Erythema(Solicited) (General disorders) | 4 (4) | 5 (8) | 2 (2) | 3 (3) | 4 (4) | 3 (3)
Vaccination Site Pain(Solicited) (General disorders) | 23 (38) | 22 (39) | 24 (34) | 19 (26) | 15 (18) | 19 (22)
Vaccination Site Swelling(Solicited) (General disorders) | 5 (7) | 7 (8) | 3 (3) | 4 (4) | 2 (2) | 4 (5)
Covid-19 (Infections and infestations) | 7 (7) | 4 (4) | 4 (4) | 4 (4) | 7 (7) | 6 (6)
Gastroenteritis (Infections and infestations) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 5 (6) | 3 (3) | 6 (10) | 2 (3) | 0 (0) | 5 (5)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 5 (7) | 2 (2) | 0 (0) | 0 (0) | 4 (6)
Myalgia(Solicited) (Musculoskeletal and connective tissue disorders) | 18 (21) | 11 (15) | 14 (18) | 13 (16) | 9 (11) | 5 (6)
Headache(Solicited) (Nervous system disorders) | 16 (28) | 20 (26) | 17 (20) | 12 (17) | 17 (21) | 16 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT05007080/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT05007080/SAP_002.pdf